CLINICAL TRIAL: NCT02952911
Title: Monitoring of Multiple Sclerosis (MS) Participants With the Use of Digital Technology (Smartphones and Smartwatches) - A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MA30162
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: MS Participants (Experimental): MS participants will perform various active tests (daily, weekly or bi-weekly) and passive monitoring (daily) using smartphone and smartwatch over 24 weeks.
  Interventions: Device: Smartphone and Smartwatch
- B: Healthy Controls (Other): Healthy participants will perform various active tests (daily, weekly or bi-weekly) and passive monitoring (daily) using smartphone and smartwatch over 24 weeks.
  Interventions: Device: Smartphone and Smartwatch

INTERVENTIONS:
Device: Smartphone and Smartwatch — Multiple sclerosis participants and healthy controls are required to wear the smartwatch; and to carry smartphone preferably in a median position in a belt bag, or alternatively in their pocket as they go about their daily routine.

SUMMARY:
This prospective pilot study will assess the feasibility of remote participant monitoring using digital technology in participants with MS and healthy controls. At the enrollment visit, the participants as well as the healthy controls will be provided with a remote patient monitoring solution which includes preconfigured smartphone and smartwatch. The configured smartphone and smartwatch pair will contain application software that prompts the user to perform various assessments, referred to as active tests and passive monitoring. Active tests will include Hand Motor Function Test (HMFT), gait test, static balance test, electronic version of the Symbol Digit Modalities Test (eSDMT), Mood Scale Question (MSQ), MS Impact Scale (29-item scale) (MSIS-29) questionnaire, MS Symptom Tracking (MSST). Passive monitoring will be done to collect metrics on gait and mobility throughout the daily life of participants in a continuous and unobtrusive manner.

ELIGIBILITY:
Inclusion Criteria:

For MS Participants:

* Definite diagnosis of MS, confirmed as per the revised McDonald 2010 criteria
* Expanded Disability Status Scale (EDSS) of 0.0 to 5.5, inclusive

For All Participants:

* Weight: 45 to 110 kilograms (kg)

Exclusion Criteria:

For MS Participants:

* Severely ill and unstable participants as per investigator's discretion
* Change in dosing regimen or switch of Disease Modifying Therapy (DMT) in the last 12 weeks prior to enrollment

For All Participants:

* Pregnant or lactating, or intending to become pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Compliance Level: Number of Active and Passive Tests Conducted by MS Participants and Healthy Controls in 12 Weeks | Week 12
Compliance Level: Number of Active and Passive Tests Conducted by MS Participants and Healthy Controls in 24 Weeks | Week 24
Satisfaction Questionnaire Score at Week 12: Assessment of MS Participants' and Healthy Volunteers' Experience Regarding Smartphone and Smartwatch Use and its Impact on Their Daily Activities | Week 12
Satisfaction Questionnaire Score at Week 24: Assessment of MS Participants' and Healthy Volunteers' Experience Regarding Smartphone and Smartwatch Use and its Impact on Their Daily Activities | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- UCSF- Multiple Sclerosis Centre; Department of Neurology, San Francisco, California, United States
- Hospital Vall d'Hebron; Servicio de Neurología, Barcelona, Spain

REFERENCES:
- [Derived] Graves JS, Elantkowski M, Zhang YP, Dondelinger F, Lipsmeier F, Bernasconi C, Montalban X, Midaglia L, Lindemann M. Assessment of Upper Extremity Function in Multiple Sclerosis: Feasibility of a Digital Pinching Test. JMIR Form Res. 2023 Oct 2;7:e46521. doi: 10.2196/46521. PMID 37782540
- [Derived] Montalban X, Graves J, Midaglia L, Mulero P, Julian L, Baker M, Schadrack J, Gossens C, Ganzetti M, Scotland A, Lipsmeier F, van Beek J, Bernasconi C, Belachew S, Lindemann M, Hauser SL. A smartphone sensor-based digital outcome assessment of multiple sclerosis. Mult Scler. 2022 Apr;28(4):654-664. doi: 10.1177/13524585211028561. Epub 2021 Jul 14. PMID 34259588
- [Derived] Midaglia L, Mulero P, Montalban X, Graves J, Hauser SL, Julian L, Baker M, Schadrack J, Gossens C, Scotland A, Lipsmeier F, van Beek J, Bernasconi C, Belachew S, Lindemann M. Adherence and Satisfaction of Smartphone- and Smartwatch-Based Remote Active Testing and Passive Monitoring in People With Multiple Sclerosis: Nonrandomized Interventional Feasibility Study. J Med Internet Res. 2019 Aug 30;21(8):e14863. doi: 10.2196/14863. PMID 31471961